CLINICAL TRIAL: NCT07196657
Title: Comparing the Efficacy and Safety of Pregabalin Monotherapy Versus Other Neuromodulatory Drugs (Crisugabalin) in the Treatment of Fibromyalgia: A Multicenter Clinical Study
Brief Title: The Efficacy and Safety of Pregabalin and Crisugabalin in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Peking University Third Hospital (Other); The Fourth Affiliated Hospital of Harbin Medical University (Other); Zhongnan Hospital (Other); Xiangya Hospital of Central South University (Other); The Affiliated Hospital of Yanbian University (Other); The Second Hospital University of South China (Other); First Affiliated Hospital of Lanzhou University (Unknown)
Responsible Party: Principal Investigator, Fang Luo, Director, Department of Pain Management, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-217-03-02
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia; Pregabalin; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin group (Active Comparator)
  Interventions: Drug: Pregabalin
- Crisugabalin group (Experimental)
  Interventions: Drug: Crisugabalin

INTERVENTIONS:
Drug: Pregabalin — For the pregabalin group, treatment will be initiated at a dosage of 150 mg daily, administered into 2 or 3 divided doses. After 3 to 7 days, the dose will be titrated to 300 mg per day, with subsequent incremental increases of 150 mg daily permitted at 3-day to 7-day intervals based on therapeutic response and tolerability, up to a maximum dose of 450 mg daily.
  Arms: Pregabalin group
Drug: Crisugabalin — For the crisugabalin group, therapy will begin at 20 mg twice daily, with a maximum allowable dose of 40 mg twice daily.
  Arms: Crisugabalin group

SUMMARY:
Fibromyalgia (FM) is a chronic pain syndrome characterized by widespread pain, fatigue, and emotional disorders. Its onset is related to factors such as central sensitization and imbalance of neurotransmitters. The current mainstream treatments include pregabalin, but the efficacy of pregabalin is limited, with only 25%-40% pain relief rate, and adverse reactions are common. crisugabalin, a new highly selective α2δ ligand, has shown potential in animal models or preliminary clinical trials, but there is insufficient evidence for its application in FM. This study aims to explore the effectiveness and safety of pregabalin or crisugabalin in treating FM, with the aim of providing a better treatment option for FM patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FM according to the 2016 Revisions to the 2010/2011 FM diagnostic criteria;
* Aged over 18 years old;
* Suffering from moderate to severe FM, refractory to non-pharmacological interventions and without prior exposure to recommend pharmacological treatments for FM;
* Baseline numeric rating scale (NRS) score of 4 or higher;
* Aspartate aminotransferase and alanine aminotransferase levels below twice the upper limit of normal range;
* Estimated glomerular filtration rate (eGFR) of at least 30 mL/min/1.73 m²;
* Willingness to provide informed consent and adequate cognitive and language capabilities to meet all study requirements;

Exclusion Criteria:

* Previous allergic reactions to pregabalin, crisugabalin, or any of their excipients;
* Prior diagnosis of epilepsy or depression requiring antidepressant therapy;
* Women who are pregnant or breastfeeding;
* Has severe systemic illnesses, such as poorly controlled hypertension, poorly controlled diabetes mellitus, or significant cardiac impairment;
* Suffering from acute or chronic pain disorders other than FM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving pain relief | At the 12-weeks
  The proportion of patients achieving pain relief defined as the proportion of patients whose baseline average pain intensity is reduced by at least 50%. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.

SECONDARY OUTCOMES:
The average pain intensity | At the weeks 1, 2, 4, 8, and 12
  The average pain intensity. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
The worst pain intensity | At the weeks 1, 2, 4, 8, and 12
  The worst pain intensity. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
Dose of crisugabalin or pregabalin | At the week 1, 2, 4, 8, 12
  the dose of experimental drug
Average weekly consumption of rescue analgesics | at weeks 4, 8, 12
  Acetaminophen will be permitted as rescue medication for FM-related pain, at doses up to 1000 mg per administration and not exceeding 3000 mg per day. All rescue medication use, including dose and frequency, will be recorded prospectively.
The Revised FM Impact Questionnaire | At the weeks 4, 8, and 12
  The Revised FM Impact Questionnaire is a 21-item self-administered questionnaire, based on symptoms reported within the preceding 7 days. The total score ranges from 0 to 100, with higher values indicating worse health status.
The Brief Pain Inventory (BPI) severity (BPI-S) and interfere (BPI-I) subsc | At the weeks 4, 8, and 12
  The BPI-S assesses pain intensity over the past 24 hours, including 4 items. The BPI-I evaluates the degree to which pain interferes with daily activities, comprising 7 items. Each BPI item is rated on a 0 to 10 NRS, with 0 represents no pain or does not interfere, and 10 represents worst pain imaginable or interferes completely. Higher scores indicate greater pain severity or interfere.
The short-form 36 Health Survey (SF-36) | At the weeks 4, 8, and 12
  The SF-36 assesses health-related quality of life, capturing preferences across various health states. It assesses 8 dimensions: physical functioning, physical role limitations due to physical health, bodily pain, general health, vitality, social functioning, emotional role limitations due to emotional problems, and mental health. Scores range from 0 to 100 for each dimension, with higher scores indicating better health status.
Patient Global Impression of Change Scale | at week 12
  A 7-point patient-reported Likert scale for evaluating subjective overall change in health/symptoms from baseline, used to assess treatment efficacy in clinical research and practice.
The Medical Outcomes Study Sleep Scale (MOS) | At the weeks 4, 8, and 12
  The MOS uses a 6-point scale to evaluate various dimensions of sleep, consisting of 12 items. A score of 1 indicates persistent presence, with a score of 6 denotes complete absence.
The Beck Depression Inventory-Ⅱ (BD-Ⅱ) | At the weeks 4, 8, and 12
  The BD-Ⅱ employs a 4-point scale (ranging from 0 to 3) to evaluate the severity of depressive symptoms, comprising 21 items in total. A score of 0 indicates the absence of symptoms, while a score of 3 reflects severe symptomatology.
Adverse Events | Through study completion, an average of 12 weeks
  Adverse Events are defined as events that occur the course of treatment, were not present before prior to the intervention, or represent a worsening of pre-existing conditions. These events will be systematically documented and categorized by severity into grades such as mild, moderate, severe, or life-threatening.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing 100070, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- See also: Mathieson S, Lin C-WC, Underwood M, Eldabe S. Pregabalin and gabapentin for pain. BMJ. 2020;369:m1315. doi: 10.1136/bmj.m1315 — https://pubmed.ncbi.nlm.nih.gov/32345589/
- See also: Domon Y, Arakawa N, Inoue T, Matsuda F, Takahashi M, Yamamura N, et al. Binding Characteristics and Analgesic Effects of Mirogabalin, a Novel Ligand for the α2δ Subunit of Voltage-Gated Calcium Channels. J Pharmacol Exp Ther. 2018;365(3):573-82. doi: 10. — https://pubmed.ncbi.nlm.nih.gov/29563324/
- See also: Gou X, Yu X, Bai D, Tan B, Cao P, Qian M, et al. Pharmacology and Mechanism of Action of HSK16149, a Selective Ligand of α2δ Subunit of Voltage-Gated Calcium Channel with Analgesic Activity in Animal Models of Chronic Pain. J Pharmacol Exp Ther. 2021;376 — https://pubmed.ncbi.nlm.nih.gov/33293377/
- See also: Chen Q, Wu Q, Song R, Wang Y, Zhang M, Li F, et al. A phase I study to evaluate the safety, tolerability, and pharmacokinetics of a novel, potent GABA analog HSK16149 in healthy Chinese subjects. Front Pharmacol. 2023;14:1296672. — https://pubmed.ncbi.nlm.nih.gov/38146463/